CLINICAL TRIAL: NCT03817853
Title: A Multicentric, Open-Label, Single Arm Study of Obinutuzumab Short Duration Infusion (SDI) in Patients With Previously Untreated Advanced Follicular Lymphoma
Brief Title: An Open-Label, Single Arm Study of Obinutuzumab Short Duration Infusion in Patients With Previously Untreated Advanced Follicular Lymphoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MO40597; 2018-003255-38 (EudraCT Number)
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Results first posted 2021-08-24 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Advanced Follicular Lymphoma
MeSH Terms: interventions — obinutuzumab; Bendamustine Hydrochloride; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Obinutuzumab+Chemotherapy (Experimental): Participants received 6-8 cycles of obinutuzumab, combined with 6 or 8 cycles of standard chemotherapy (cyclophosphamide, doxorubicin, vincristine, and prednisone/prednisolone/methylprednisolone [CHOP - 21-day cycle) or bendamustine (28-day cycle), or cyclophosphamide, vincristine, and prednisone/prednisolone/methylprednisolone [CVP - 21-day cycle]). Participants received an additional two doses of obinutuzumab on Days 8 and 15 of Cycle 1. The investigator is free to choose the chemotherapy for each patient. Obinutuzumab and chemotherapy is administered during induction phase and obinutuzumab monotherapy is administered during maintenance phase.
  Interventions: Drug: Obinutuzumab; Drug: Bendamustine; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone/Prednisolone/Methylprednisolone; Drug: Vincristine

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab 1000 mg IV infusion, administered on Day 1, 8 and 15 during Cycle 1, and on Day 1 of subsequent cycles, for 6-8 cycles. Each cycle is 21 or 28 days long depending on the chemotherapy regimen allocated. Maintenance obinutuzumab monotherapy in patients who achieve at least a partial response, after induction therapy will be administered a dose of 1000 mg once every 8 weeks for 2 years or until disease progression (whichever occurs first).
  Other Names: GA101, RO5072759
Drug: Bendamustine — Bendamustine will be administered on Days 1 and 2 for Cycles 1-6 at a dose of 90 mg/m2/day, for six 28-day cycles.
Drug: Cyclophosphamide — Cyclophosphamide 750 milligrams per square metre (mg/m^2), administered intravenously (IV) on Day 1 of each 21-day cycle, for six cycles for CHOP treatment or eight cycles for CVP treatment.
Drug: Doxorubicin — Doxorubicin 50 mg/m^2 IV, administered on Day 1 of each 21-day cycle, for six cycles.
Drug: Prednisone/Prednisolone/Methylprednisolone — Prednisone 100 mg (or equivalent prednisolone or methylprednisolone), administered orally on Days 1-5 of each 21-day cycle, for six cycles for CHOP treatment or eight cycles for CVP treatment.
Drug: Vincristine — Vincristine 1.4 mg/m^2 (maximum 2 mg) IV, administered on Day 1 of each 21-day cycle, for six cycles for CHOP treatment or eight cycles for CVP treatment.

SUMMARY:
This open-label, single arm study will evaluate the safety of obinutuzumab administered as a short duration infusion (SDI; target 90-minute infusion) during cycle 2 and from cycle 2 onwards in combination with chemotherapy in participants with previously untreated advanced follicular lymphoma (FL). The study has two phases: in the first phase, participants will receive the first cycle of obinutuzumab-based chemotherapy (G-chemo) induction therapy as usual with the first three infusions of obinutuzumab (1000 mg) administered at the regular infusion rate on Day 1, 8, and 15 of cycle 1. Phase 2 starts when participants who do not experience any Grade ≥ 3 infusion related reactions during the first cycle receive their first obintuzumab infusion given at the faster infusion rate in Cycle 2. For Cycle 2, Day 1 and all other following infusions (including maintenance), obinutuzumab will be administered at a faster infusion of 90-minute SDI, as long as the participant does not experience any Grade ≥ 3 infusion related reactions. The investigator is free to choose the chemotherapy for each participant (bendamustine, CHOP [cyclophosphamide, doxorubicin, vincristine, prednisone/prednisolone/methylprednisolone], or CVP [cyclophosphamide, vincristine, and prednisone/prednisolone/methylprednisolone]). The total number of cycles of G-chemo induction therapy and the cycles length depends on the chemotherapy chosen for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously untreated Stage III or IV FL or Stage II bulky disease scheduled to receive obinutuzumab plus chemotherapy due to at least one of the following criteria: a.) Bulky disease, defined as a nodal or extranodal (except spleen) mass

  ≥ 7 cm in the greatest diameter b.) Local symptoms or compromise of normal organ function due to progressive nodal disease or extranodal tumor mass c.) Presence of B symptoms (fever [> 38ºC], drenching night sweats, or unintentional weight loss of > 10% of normal body weight over a period of 6 months or less) d.) Presence of symptomatic extranodal disease (e.g., pleural effusions, peritoneal ascites) e.) Cytopenias due to underlying lymphoma (i.e., absolute neutrophil count < 1.0 × 109/L, hemoglobin < 10 g/dL, and/or platelet count < 100 × 109/L) f.) Involvement of ≥ 3 nodal sites, each with a diameter of ≥ 3 cm g.) Symptomatic splenic enlargement
* Histologically documented CD-20-positive FL, as determined by the local laboratory
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate hematologic function (unless abnormalities are related to FL)
* Life expectancy of ≥ 12 months
* For women who are not postmenopausal (≥ 12 consecutive months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 18 months after the last dose of obinutuzumab, for at least 3 months after the last dose of bendamustine or according to institutional guidelines for CHOP or CVP chemotherapy, whichever is longer
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures and agreement to refrain from donating sperm

Exclusion Criteria:

* Relapsed / refractory FL
* Prior treatment for FL with chemotherapy, radiotherapy, or immunotherapy
* Grade IIIb FL
* Histological evidence of transformation of FL into high-grade B-cell NHL
* Treatment with systemic immunosuppressive medications, including, but not limited to, prednisone/prednisolone/methylprednisolone (at a dose equivalent to >30 mg/day prednisone), azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents within 2 weeks prior to Day 1 of Cycle 1
* History of solid organ transplantation
* History of anti-CD20 antibody therapy
* History of severe allergic or anaphylactic reaction to humanized, chimeric, or murine monoclonal antibodies
* Known sensitivity or allergy to murine products
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any of the study drugs
* Active bacterial, viral, fungal, or other infection or any major episode of infection requiring treatment with IV antibiotics within 4 weeks of Day 1 of Cycle 1
* Positive test results for chronic HBV infection (defined as positive HBsAg serology)
* Positive test results for hepatitis C (hepatitis C virus [HCV] antibody serology testing)
* Known history of HIV positive status
* History of progressive multifocal leukoencephalopathy (PML)
* Vaccination with a live virus vaccine within 28 days prior to Day 1 of Cycle 1 or anticipation that such a live, attenuated vaccine will be required during the study
* History of prior other malignancy with the exception of: a. Curatively treated carcinoma in situ of the cervix, good-prognosis ductal carcinoma in situ of the breast, basal- or squamous-cell skin cancer, Stage I melanoma, or low-grade, early-stage localized prostate cancer b. Any previously treated malignancy that has been in remission without treatment for ≥ 2 years prior to enrollment
* Evidence of any significant, uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the previous 6 months, unstable arrhythmia, or unstable angina) or significant pulmonary disease (such as obstructive pulmonary disease or history of bronchospasm)
* Major surgical procedure other than for diagnosis within 28 days prior to Day 1 of Cycle 1, Day 1, or anticipation of a major surgical procedure during the course of the study
* Any of the following abnormal laboratory values:

  1. Creatinine > 1.5 × the upper limit of normal (ULN) (unless creatinine clearance normal) or creatinine clearance < 40 mL/min
  2. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 × ULN
  3. Total bilirubin ≥ 1.5 × the ULN: Patients with documented Gilbert disease may be enrolled if total bilirubin is ≤ 3.0 × the ULN.
  4. International normalized ratio (INR) > 1.5 in the absence of therapeutic anticoagulation
  5. Partial thromboplastin time or activated partial thromboplastin time > 1.5 × ULN in the absence of a lupus anticoagulant
* For patients who will be receiving CHOP: left ventricular ejection fraction (LVEF) < 50% by multigated acquisition (MUGA) scan or echocardiogram
* Pregnant or lactating, or intending to become pregnant during the study
* Any investigational therapy within 28 days prior to the start of Cycle 1
* Positive test results for human T-lymphotropic virus 1 (HTLV-1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-08-04 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (33):
- United States (7):
  - Rocky Mountain Cancer Center; Medical Oncology, Boulder, Colorado
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Summit Medical Center, Florham Park, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Willamette Valley Cancer Ctr - 520 Country Club, Eugene, Oregon
  - Texas Onc-Central Austin CA Ct, Austin, Texas
  - Texas Oncology Cancer Center, Austin, Texas
- Brazil (3):
  - NOHC - Núcleo de Oncologia e Hematologia do Ceará, Fortaleza, Ceará
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Amaral Carvalho, Jaú, São Paulo
- Germany (7):
  - Klinikum Chemnitz gGmbH, Klinik für Innere Medizin III, Hämatologie und Onkologie, Chemnitz
  - Klinik der Uni zu Köln; I. Med. Klinik, Cologne
  - Städtisches Klinikum Dessau, Dessau
  - Universitätsklinikum Frankfurt; Medizinische Klinik II; Onkologie, Frankfurt
  - OncoResearch Lerchenfeld GmbH, Hamburg
  - MVZ Dr. Vehling-Kaiser GmbH; Onkologische Praxis, Landshut
  - Onkologische Schwerpunktpraxis Lübeck, Lübeck
- Japan (6):
  - Chiba Cancer Center, Chiba
  - Hokkaido University Hospital, Hokkaido
  - Kobe City Medical Center General Hospital, Hyōgo
  - Kindai University Hospital, Osaka
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
- Netherlands (2):
  - Albert Schweitzer Ziekenhuis - loc Dordrecht, Dordrecht
  - Martini Ziekenhuis, Groningen
- Spain (5):
  - Hospital De Txagorritxu; Servicio de Hematologia, Vitoria-Gasteiz, Alava
  - Hospital Universitario Puerta del Mar; Servicio de Hematologia, Cadiz, Cadiz
  - Hospital del Mar; Servicio de Hematologia, Barcelona
  - Hospital Universitario la Paz; Servicio de Hematologia, Madrid
  - Hospital General Universitario J.M Morales Meseguer; Servicio de Hematología, Murcia
- United Kingdom (3):
  - University Hospital of Wales, Cardiff
  - Portsmouth Hospitals NHS Trust - Queen Alexandra Hospital, Portsmouth
  - Royal Cornwall Hospital, Truro

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 35 sites across 7 countries.
Pre-assignment Details: Of the all participants population (114 participants), one participant did not receive the study treatment, thus the safety-evaluable population included 113 participants.
Groups:
- All Participants: Participants were enrolled in an induction phase and received 6-8 cycles of obinutuzumab, combined with 6 or 8 cycles of standard chemotherapy (cyclophosphamide, doxorubicin, vincristine, and prednisone/prednisolone/methylprednisolone [CHOP - 21-day cycle) or bendamustine (28-day cycle), or cyclophosphamide, vincristine, and prednisone/prednisolone/methylprednisolone [CVP - 21-day cycle]). Participants received an additional two doses of obinutuzumab on Days 8 and 15 of Cycle 1. The investigator was free to choose the chemotherapy for each participant.
- Maintenance: Participants who achieved a partial response (PR) or complete response (CR) following the induction phase received obinutuzumab maintenance therapy. 1000 mg of obinutuzumab as single agent was administered as an SDI every 8 weeks (+ or - 10 days) for 2 years or until disease progression).
- Follow-up: Participants with stable disease (SD) or progressive disease (PD) as best response after induction therapy discontinued study treatment and underwent a safety follow-up visit at 3 months (90 days (+ or - 10 days)). All participants were followed up at 3 months (90 days (+ or - 10 days)) from the time of the last dose of study treatment.
Period: Induction Phase
Arm/Group | All Participants | Maintenance | Follow-up
Started | 113 | 0 | 0
Completed | 93 | 0 | 0
Not Completed | 20 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0
Not completed — Measures due to covid19; transformation to double hit high-grade b lymphoma; discontinuation of trt. | 3 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Progressive Disease | 6 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0
Period: Maintenance Phase
Arm/Group | All Participants | Maintenance | Follow-up
Started | 0 | 95 (3 participants started the maintenance phase after discontinuing from the induction phase due to COVID-19 measures.) | 0
Completed | 0 | 67 | 0
Not Completed | 0 | 28 | 0
Not completed — Adverse Event | 0 | 8 | 0
Not completed — Death | 0 | 5 | 0
Not completed — Progressive Disease | 0 | 7 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Various reasons | 0 | 4 | 0
Not completed — Protocol Deviation | 0 | 1 | 0
Period: Follow-up Phase
Arm/Group | All Participants | Maintenance | Follow-up
Started | 0 | 0 | 99 (14 participants discontinued the induction phase but started the follow-up phase. Note that it was not a requirement to complete the maintenance phase to be allowed to enter the follow-up phase.)
Completed | 0 | 0 | 92
Not Completed | 0 | 0 | 7
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Death | 0 | 0 | 1
Not completed — Progressive Disease | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The all participants population includes all enrolled participants.
Arm/Group | All Participants
Number analyzed (Participants) | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 57
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    Asian | 27
    White | 82
    Other | 2
    Multiple | 2
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnicity
  Participants
    Hispanic or Latino | 33
    Not Hispanic or Latino | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Grade >=3 Infusion-Related Reactions (IRRs) During Cycle 2 in Patients Who Had Previously Received Obinutuzumab at the Standard Infusion Rate During Cycle 1 Without Experiencing a Grade 3 or 4 IRR
Description: IRRs were defined as all adverse events (AEs) that occurred during or within 24 hours from the end of study treatment infusion and were judged as related to infusion of study treatment components by the investigator.
Time Frame: Within 24 hours from the end of study treatment infusion of Day 1 in Cycle 2 (1 cycle: 21 or 28 days depending on the chemotherapy selected)
Population: The Short Duration Infusion (SDI) population included all enrolled particpants who did not experience a Grade 3 or 4 IRR during cycle 1 (i.e. at any of the three Cycle 1 infusions), received obinutuzumab given at the standard rate only during Cycle 1, and received obinutuzumab as an SDI at cycle 2.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | All Participants
Number analyzed (Participants) | 99
Percentage of Participants | 0 [0.00 to 3.66]

2. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant who was administered a pharmaceutical product, regardless of causal attribution. An AE was therefore any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Pre-existing conditions which worsened during the study, recurrence of an intermittent medical condition, deterioration in a laboratory value or other clinical test or were related to a protocol-mandated intervention were also considered AEs. Grading was completed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0.
Time Frame: Baseline up to end of study (approximately 4 years)
Population: The safety population included all participants who received at least one dose of obinutuzumab.
Measure: Number; unit: Percentage of Participants
Groups:
- Maintenance: Obinutuzumab: Participants received 6-8 cycles of obinutuzumab, combined with 6 or 8 cycles of standard chemotherapy (cyclophosphamide, doxorubicin, vincristine, and prednisone/prednisolone/methylprednisolone [CHOP - 21-day cycle) or bendamustine (28-day cycle), or cyclophosphamide, vincristine, and prednisone/prednisolone/methylprednisolone [CVP - 21-day cycle]). Participants received an additional two doses of obinutuzumab on Days 8 and 15 of Cycle 1. The investigator was free to choose the chemotherapy for each participant.
  Participants who achieved a partial response (PR) or complete response (CR) following the induction phase received obinutuzumab maintenance therapy. 1000 mg of obinutuzumab as single agent was administered as an SDI every 8 weeks (+ or - 10 days) for 2 years or until disease progression).
Arm/Group | All Participants | Maintenance: Obinutuzumab | Follow-up
Number analyzed (Participants) | 113 | 95 | 99
Percentage of Participants | 99.1 | 90.5 | 27.3

3. Secondary Outcome: Percentage of IRRs Regardless of Grade by Cycle
Description: as for outcome 1
Time Frame: Within 24 hours from the end of study treatment infusion in all cycles, including maintenance ((1 cycle: 21 or 28 days depending on the chemotherapy selected); up to approximately 2.5 years)
Population: The safety population included all participants who received at least one dose of obinutuzumab.
Measure: Number; unit: Percentage of Participants
Arm/Group | All Participants
Number analyzed (Participants) | 113
Percentage of Participants
  Cycle 1 Day 1 | 50.4
  Cycle 1 Day 2: number analyzed (Participants) | 51
  Cycle 1 Day 2 | 7.8
  Cycle 1 Day 8: number analyzed (Participants) | 112
  Cycle 1 Day 8 | 5.4
  Cycle 1 Day 15: number analyzed (Participants) | 111
  Cycle 1 Day 15 | 4.5
  Cycle 2: number analyzed (Participants) | 110
  Cycle 2 | 11.8
  Cycle 3: number analyzed (Participants) | 108
  Cycle 3 | 8.3
  Cycle 4: number analyzed (Participants) | 108
  Cycle 4 | 6.5
  Cycle 5: number analyzed (Participants) | 107
  Cycle 5 | 5.6
  Cycle 6: number analyzed (Participants) | 105
  Cycle 6 | 4.8
  Cycle 7: number analyzed (Participants) | 55
  Cycle 7 | 3.6

4. Secondary Outcome: Time to IRR From Infusion to Onset of the IRR During Cycle 2
Description: Time to IRR (of any grade) in Cycle 2 was defined as the time from the start of infusion (i.e., start date/time of infusion of the first component of study treatment) in Cycle 2 to the onset of the IRR (of any grade) during Cycle 2.
Time Frame: From infusion to onset of IRR during Cycle 2 (1 cycle: 21 or 28 days depending on the chemotherapy selected)
Population: The SDI population included all enrolled participants who did not experience a Grade 3 or 4 IRR during cycle 1 (i.e. at any of the three Cycle 1 infusions), received obinutuzumab given at the standard rate only during Cycle 1, and received obinutuzumab as an SDI at cycle 2. For this outcome measure, only one participant was analyzed.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | All Participants
Number analyzed (Participants) | 1
Hours | 11.800 (NA) — Standard deviation (SD) is not available because only 1 participant had the time to IRR recorded and the SD for one value is not defined.

5. Secondary Outcome: Duration (In Minutes) of Obinutuzumab Administration by Cycle
Description: The duration of obinutuzumab administration (in minutes) by cycle was defined as the difference between the end time and the start time of obinutuzumab administration.
Time Frame: All cycles including maintenance (1 cycle: 21 or 28 days depending on the chemotherapy selected; up to approximately 2.5 years)
Population: The safety population included all participants who received at least one dose of obinutuzumab.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | All Participants
Number analyzed (Participants) | 113
Minutes
  Cycle(C) 1 Day(D) 1: number analyzed (Participants) | 100
  Cycle(C) 1 Day(D) 1 | 295.96 (147.87)
  C1D8: number analyzed (Participants) | 107
  C1D8 | 215.97 (46.99)
  C1D15: number analyzed (Participants) | 102
  C1D15 | 208.91 (33.13)
  C2: number analyzed (Participants) | 103
  C2 | 99.61 (13.36)
  C3: number analyzed (Participants) | 101
  C3 | 103.29 (65.45)
  C4: number analyzed (Participants) | 101
  C4 | 99.26 (13.90)
  C5: number analyzed (Participants) | 100
  C5 | 98.46 (16.48)
  C6: number analyzed (Participants) | 102
  C6 | 99.10 (12.18)
  C7: number analyzed (Participants) | 51
  C7 | 98.84 (13.61)
  C8: number analyzed (Participants) | 50
  C8 | 95.68 (4.12)
  Maintenance Week 1: number analyzed (Participants) | 83
  Maintenance Week 1 | 97.64 (10.08)
  Maintenance Week 9: number analyzed (Participants) | 63
  Maintenance Week 9 | 96.78 (8.49)
  Maintenance Week 17: number analyzed (Participants) | 48
  Maintenance Week 17 | 97.77 (7.66)
  Maintenance Week 25: number analyzed (Participants) | 31
  Maintenance Week 25 | 97.16 (7.23)
  Maintenance Week 33: number analyzed (Participants) | 24
  Maintenance Week 33 | 95.08 (4.27)
  Maintenance Week 41: number analyzed (Participants) | 13
  Maintenance Week 41 | 95.77 (5.26)
  Maintenance Week 49: number analyzed (Participants) | 9
  Maintenance Week 49 | 93.56 (4.48)
  Maintenance Week 57: number analyzed (Participants) | 2
  Maintenance Week 57 | 93.50 (4.95)

6. Secondary Outcome: Type of Grade >=3 IRRs Associated With the Obinutuzumab Administered as an SDI by Cycle
Time Frame: as for outcome 5
Population: The safety population included all participants who received at least one dose of obinutuzumab. Only 1 participant had a Grade >=3 IRR, with 3 symptoms in Cycle 5. Weight increased was a grade 1 symptom belonging to the grade 3 IRRs.
Measure: Number; unit: Percentage of Participants
Arm/Group | All Participants
Number analyzed (Participants) | 113
Percentage of Participants
  Cycle (C) 5- Hypertension: number analyzed (Participants) | 1
  Cycle (C) 5- Hypertension | 33.3
  C5 - Renal failure: number analyzed (Participants) | 1
  C5 - Renal failure | 33.3
  C5 - Weight increased: number analyzed (Participants) | 1
  C5 - Weight increased | 33.3

7. Secondary Outcome: Duration of Grade >=3 IRRs Associated With the Obinutuzumab Administered as an SDI by Cycle
Description: The duration, in minutes, of IRRs during all cycles, where obinutuzumab was administered as an SDI.
Time Frame: as for outcome 5
Population: The safety population (113 participants) included all participants who received at least one dose of obinutuzumab.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | All Participants
Number analyzed (Participants) | 1
Minutes | 165.0 (NA) — SD is not available because only 1 participant had the duration of IRR recorded and the SD for one value is not defined.

8. Secondary Outcome: Objective Response Rate (ORR) at the End of Induction (EOI) Therapy
Description: ORR at EOI therapy was defined as the percentage of particpants with either a CR, CR unconfirmed or PR at the EOI visit, as determined by the investigator and according to the guidelines used at the site.
Time Frame: Baseline up to end of induction therapy (up to approximately 6 months)
Population: The safety population included all participants who received at least one dose of obinutuzumab.
Measure: Number; unit: Percentage of Participants
Arm/Group | All Participants
Number analyzed (Participants) | 113
Percentage of Participants
  Complete Response: number analyzed (Participants) | 77
  Complete Response | 68.1
  Complete Response unconfirmed: number analyzed (Participants) | 0
  Partial Response: number analyzed (Participants) | 22
  Partial Response | 19.5

9. Secondary Outcome: Progression-Free Survival (PFS) Rate at the End of the Study
Description: PFS was defined as the time from start of treatment to the first occurrence of disease progression as assessed by the investigator according to the guidelines used at the site or death from any cause.
Time Frame: Baseline up to end of study (up to approximately 4 years)
Population: The safety population included all participants who received at least one dose of obinutuzumab.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Participants
Number analyzed (Participants) | 113
Months | 33.97 [32.13 to NA] — Due to the low number of events, the upper CI limit was not evaluable.

10. Secondary Outcome: Overall Survival (OS) at the End of the Study
Description: OS was defined as the time from start of treatment (date of first intake of any study treatment component) to death from any cause.
Time Frame: Baseline up to end of study (up to approximately 4 years)
Population: The safety population included all participants who received at least one dose of obinutuzumab.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Participants
Number analyzed (Participants) | 113
Months | NA [33.97 to NA] — The median could not be estimated due to the low number of events.

11. Secondary Outcome: Complete Response (CR) Rate at 30 Months (CR30), as Assessed by the Investigator and According to the Guidelines Used at the Site
Description: The CR30 rate was defined as the percentage of participants with a CR at 30 months from study treatment initiation (date of first intake of any study treatment component), as determined by the investigator according to the guidelines used at the site.
Time Frame: Baseline up to 30 months
Population: The safety population included all participants who received at least one dose of obinutuzumab.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | All Participants
Number analyzed (Participants) | 113
Percentage of Participants | 55.6 [45.68 to 65.12]

ADVERSE EVENTS:
Time Frame: Baseline up to end of study (approximately 4 years)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant who was administered a pharmaceutical product, regardless of causal attribution. Grading was completed according to the CTCAE, version 5.0.
Arm/Group | All Participants | Maintenance | Follow-up
All-Cause Mortality (participants affected / at risk) | 9/113 | 8/95 | 4/99
Serious Adverse Events (participants affected / at risk) | 21/113 | 17/95 | 11/99
Other Adverse Events (participants affected / at risk) | 111/113 | 76/95 | 13/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=113) | Maintenance (N=95) | Follow-up (N=99)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 4 (4)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 2 (3) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 4 (4) | 3 (3)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Severe acute respiratory syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=113) | Maintenance (N=95) | Follow-up (N=99)
Anaemia (Blood and lymphatic system disorders) | 20 (25) | 3 (3) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 20 (34) | 3 (6) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 22 (36) | 4 (5) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 68 (116) | 16 (27) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 20 (28) | 4 (8) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 11 (13) | 3 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 9 (10) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 39 (42) | 6 (6) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 15 (18) | 5 (6) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 8 (8) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 48 (67) | 4 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 15 (17) | 1 (1) | 0 (0)
Asthenia (General disorders) | 11 (13) | 6 (6) | 1 (1)
Fatigue (General disorders) | 18 (19) | 3 (3) | 1 (1)
Malaise (General disorders) | 12 (15) | 2 (2) | 0 (0)
Mucosal inflammation (General disorders) | 9 (9) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 15 (18) | 11 (14) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 2 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 6 (7) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 69 (128) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 10 (14) | 4 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 7 (10) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 3 (3) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 7 (7) | 5 (6) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (16) | 8 (9) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 11 (14) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 7 (7) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 18 (19) | 7 (7) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 19 (19) | 3 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (13) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 19 (19) | 5 (5) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 12 (13) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 17 (18) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (7) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 7 (8) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 5 (5) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 4 (4) | 4 (4) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 11 (12) | 5 (5)
Herpes zoster (Infections and infestations) | 4 (4) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (4) | 6 (6) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 6 (7) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 4 (4) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2) | 8 (8) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 13 (14) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 0 (0)
Paraesthesia (Nervous system disorders) | 5 (5) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 6 (6) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (5) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 7 (8) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT03817853/Prot_002.pdf
  • Statistical Analysis Plan (2020-07-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT03817853/SAP_001.pdf